CLINICAL TRIAL: NCT05977738
Title: Phase 0 lead-in Trial of Pitavastatin in Primary and Recurrent Glioblastoma Patients
Brief Title: Repurposed Drugs in Research for Cancer Clinical Trials- Pitavastatin
Acronym: ReDiReCCT-Pita
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: C.Dirven (Other)
Responsible Party: Sponsor-Investigator, C.Dirven, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2023-505743-38-00; UTN U1111-1294-4392 (Other: WHO)
Record Dates: First submitted 2023-07-25; First posted 2023-08-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma Multiforme, Adult; Recurrent Glioblastoma
Keywords: Phase 0; GBM; Glioma; Pitavastatin
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — pitavastatin

STUDY DESIGN:
Intervention Model Description: open label, dose-finding, 3+3-like dose-escalation study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose group 1: 16 mg (Experimental): Pitavastatin 16 mg via oral route in the form of daily tablets for 6 days before SOC surgery
  Interventions: Drug: Pitavastatin calcium
- Dose group 2: 32 mg (Experimental): Pitavastatin 32 mg via oral route in the form of daily tablets for 6 days before SOC surgery
  Interventions: Drug: Pitavastatin calcium
- Dose group 3: 48 mg (Experimental): Pitavastatin 48 mg via oral route in the form of daily tablets for 6 days before SOC surgery
  Interventions: Drug: Pitavastatin calcium

INTERVENTIONS:
Drug: Pitavastatin calcium — Daily Pitavastatin administration
  Other Names: Alipza

SUMMARY:
The goal of this Phase 0 trial is to study if pre-operative oral pitavastatin administration reaches the tumour in patients with primary or a recurrent glioblastoma. The main question[s] it aims to answer are:

* Does pitavastatin reach a cytotoxic concentration in gadolinium-enhanced tumour tissue after oral administration?
* Does pitavastatin achieve a concentration that can synergize with temozolomide in the gadolinium non-enhanced area of the tumour?

Participants will receive pitavastatin in differing dosages a week before their elective surgery and blood and tumour samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for resection of a suspected primary glioblastoma or a recurrent glioblastoma.
2. MRI- measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 1 perpendicular measurement of at least 0.5 cm.
3. Adequate Renal Function defined as: estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 by Chronic Disease Epidemiology Collaboration (CKD-EPI) equation.
4. CK elevation 3 X ULN.
5. Ability to understand and the willingness to sign a written informed consent document.
6. Participant has voluntarily agreed to participate by giving written informed consent Written informed consent for participation in the protocol must be obtained prior to any screening procedures taking place.
7. Willingness and ability to comply with all scheduled visits, treatment plans, laboratory tests and other procedures.
8. Age ≥18 years at time of consent.
9. Ability and willingness to swallow oral medication.
10. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
11. For females of reproductive potential: use of highly effective contraception method defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly.
12. Females of child-bearing potential must agree not to breastfeed starting at screening, and throughout the study period.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Known allergic reactions to components of the pitavastatin calcium tablets.
3. Patients with ALAT and ASAT levels 3 X ULN.
4. Unwillingness to temporarily stop an already prescribed statin, during treatment with pitavastatin.
5. Active infection or fever >38.5°C requiring systemic antibiotic, antifungal or antiviral therapy.
6. Concomitant use of cyclosporin, gemfibrozil, systemic fusidic acid, fibrates, niacin or colchicine.
7. Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, unexplained elevated liver transaminase levels, and active and chronic hepatitis as determined by the investigator.
8. Suspicion of oral malabsorption, influencing the uptake of drugs from the ileum, such as Morbus Crohn.
9. Treatment with another investigational drug or other intervention within 30 days prior to enrolment or within 5 half-lives of the investigational product, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Intratumoral pitavastatin concentration as assessed by LC-MS analysis on tumour tissue. | From the last patient visit of each dose cohort at day 9 to 2 weeks after the last patient visit of each dose cohort.
  Detection of pitavastatin in gadolinium enhanced and gadolinium non-enhanced tumour. tissue in relation to serum levels after preoperative administration.

SECONDARY OUTCOMES:
Tolerability of short-term pitavastatin treatment as assesseb by a customized questionnaire related to adverse events found during the use of pitavastatin. | From the last patient visit of the last dose cohort to 2 weeks after the last patient visit of the last dose cohort on day 9.
  Number of AEs, SAEs and SUSARs collected at the end of the trial. Events will be scored according to CTC criteria version 5.0 (Published November 27th, 2017).
Relation of plasma pitavastatin concentration and intratumoral pitavastatin concentration as assessed by LC-MS analysis on plasma and tumour tissue. | From the moment the LC-MS analysis of the last patient tumour tissue and plasma is performed to two weeks after the last patient visit on day 9 of the last dose cohort.
  Correlation of pitavastatin concentration in plasma to pitavastatin concentration in different tumour sites(gadolinium enhanced, gadolinium non-enhanced and tumour periphery).

OTHER OUTCOMES:
Differences in RNA expression after pitavastatin exposure in tumour tissue using RNA sequencing. | From the last tumour tissue acquisition of the last patient of the last dose cohort to 3 months after all tissue is collected.
  Using RNA sequencing on collected tumour samples from the gadolinium enhanced part of the tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Dirven, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided